CLINICAL TRIAL: NCT03229382
Title: Evaluation of Efficacy and Safety of Obinutuzumab Preemptive Treatment at the Time of the Molecular Relapse After First Line Immunochemotherapy With Autologous Stem Cell (ML29157).
Brief Title: Efficacy and Safety of Obinutuzumab Preemptive Treatment at the Time of the Molecular Relapse
Acronym: OPERA-PLRG10
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Very slow recruitment due to lack of relapse in the observed group of patients
Sponsor: Polish Lymphoma Research Group (Network)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML29157; 2015-005439-41 (EudraCT Number)
Record Dates: First submitted 2017-07-10; First posted 2017-07-25 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Mantle Cell Lymphoma
Keywords: MCL, obinutuzumab
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Obinutuzumab 1000 mg IV infusion, day: 1, 8, 15, 22 (Experimental): Patients with evidence of MCL molecular relapse defined as an increasing copy number in quantitative real-time polymerase chain reaction (RQ-PCR) of clone-specific immunoglobulin heavy chain (IGH) gene rearrangements or BCL1-IGH fusion genes according to BIOMED-2 methodology and protocols in peripheral blood or/and bone marrow without evidence of clinical relapse/progression after auto-HCT procedure with all inclusion and no exclusion clinical trial criteria will receive 4 weekly infusions of obinutuzumab.
  Interventions: Drug: Obinutuzumab

INTERVENTIONS:
Drug: Obinutuzumab — Patients, in whom all inclusion criteria have been confirmed and all exclusion criteria have been ruled out, will receive 4 intravenous infusions of obinutuzumab (GA101, Gazyvaro) at a dose of 1000 mg on Days 1, 8, 15 and 22.
  Other Names: Gazyvaro; GA101

SUMMARY:
The objective of the study is the evaluation of efficacy and safety of obinutuzumab preemptive treatment at the time of the molecular relapse after first line immunochemotherapy with autologous stem cell transplantation in mantle cell lymphoma patients.

DETAILED DESCRIPTION:
Patients with evidence of MCL molecular relapse defined as an increasing copy number in quantitative real-time polymerase chain reaction (RQ-PCR) of clone-specific immunoglobulin heavy chain (IGH) gene rearrangements or BCL1-IGH fusion genes according to BIOMED-2 methodology and protocols in peripheral blood or/and bone marrow without evidence of clinical relapse/progression after auto-HCT procedure with all inclusion and no exclusion clinical trial criteria will receive 4 weekly infusions of obinutuzumab (1000 mg, iv) on day 1, 8, 15, 22.Response assessment in bone marrow and/or peripheral blood and CT/MRI imaging will be performed 2 months after the obinutuzumab preemptive treatment. Patients with subsequent molecular remission in peripheral blood and/or bone marrow confirmed in RQ-PCR (with 10-4 level of sensitivity) assessment and no signs of relapse/progression according to the Lugano Classification will be further followed. From this moment, evaluation of response will be performed every 6 months with computed tomography/magnetic resonance (CT/MR) imaging and bone marrow aspiration to detect classical relapse/progression and/or to detect subsequent molecular relapse by quantitative real-time polymerase chain reaction (RQ-PCR) of clone-specific immunoglobulin heavy chain (IGH) gene rearrangements or BCL1-IGH fusion genes with the use of consensus JH probes and specific ASO primers. Patients will be monitored every 3 months (outpatient visits with peripheral blood samples for MRD assessment to detect molecular relapse by quantitative RQ-PCR of clone-specific immunoglobulin heavy chain (IGH) gene rearrangements or BCL1-IGH fusion genes). Preemptive treatment can be administered in subsequent molecular relapses/progressions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with evidence of MCL molecular relapse in peripheral blood or/and bone marrow,
* Diagnosis of mantle cell lymphoma confirmed by histopathology
* Presence of clone-specific immunoglobulin heavy chain (IGH) gene rearrangements or BCL1-IGH fusion gene as a molecular marker used for minimal residual disease (MRD) assessment,
* Patients in CR/PR after first-line treatment with myeloablative consolidation and ASCT,
* Patients without evidence of mantle cell lymphoma progression/relapse according to the Lugano Classification criteria (2014),
* ECOG performance status ≤ 2,
* Signed patient's informed consent form,
* Survival prognosis > 6 months,
* Women of childbearing potential must have a negative pregnancy test result prior to initiation of treatment with the study medication and must consent to undergo pregnancy tests during the treatment period.,
* Women of child-bearing potential must consent either to sexual abstinence or to using effective contraception (that results in a failure rate of < 1% per year) while receiving the study medication and for 18 months after its discontinuation,
* Men must consent either to using an acceptable contraception method (that results in a failure rate of < 1% per year) or continued sexual abstinence while receiving the study medication and for 6 months after its discontinuation.

Exclusion Criteria:

* Central nervous system involvement,
* Chemotherapy, radiation therapy or any other antineoplastic treatment (including steroids, monoclonal antibodies or medications at the stage of clinical studies, before receiving marketing authorisation) after ASCT and before administration of the study medication,
* Major surgery within 28 days prior to the study treatment initiation,
* Renal impairment (plasma creatinine concentration > 1.5 × upper limit of normal and/or creatinine clearance ≤ 40 ml/h),
* Hepatic impairment (total bilirubin concentration > 1.5 × upper limit of normal, AST and ALT > 2.5 × upper limit of normal),
* Hb< 9 g/dl, ANC < 1.5 G/l, platelets < 75 G/l,
* International normalized ratio (INR) > 1.5,
* Clinically significant heart disease, including uncontrolled arrhythmias, unstable coronary artery disease, serious congestive circulatory failure (NYHA III-IV), myocardial infarction within 6 months before enrolment,
* Other comorbidities, not responding to treatment, including, but not limited to: hematopoietic system diseases, gastrointestinal system diseases, endocrine system diseases, respiratory system diseases, neurological diseases, cerebral diseases and mental diseases that could affect compliance with the protocol or interpretation of results,
* Active infections (viral, bacterial, fungal),
* Coexistence of another neoplasm or a history of neoplastic disease (except for adequately treated basal cell carcinoma or squamous cell skin carcinoma, in situ cervical cancer or other neoplasm if the patient is in complete remission after at least 5 years of treatment discontinuation),
* Active HIV, HBV or HCV infection,
* Positive test results for chronic hepatitis B. All patients must be tested for both HBsAg and HBcAb at screening, if either of the tests is positive, the patient is not eligible for inclusion in the trial. Patients who have protective titers of HBsAb after vaccination are eligible provided they are negative for both HBsAg and HBcAb,
* Positive testing for hepatitis C (hepatitis C virus [HCV] antibody serology testing). Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA,
* Vaccination with live vaccines within 28 days prior to start of the preemptive treatment,
* Known or suspected hypersensitivity to the study medication,
* Women who are pregnant or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
MRD negativity defined as a MRD level | 2 months after obinutuzumab treatment
  Molecular response rate (molRR) defined as a rate of molecular response with at least 10-4 sensitivity level assessed by quantitative RQ-PCR

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 3 years and 2 month
  defined as the time from the date of the first obinutuzumab infusion to disease progression or relapse, as determined by the investigator using the Lugano Classification or death from any cause after the last dose of study drug
Time to molecular relapse | 3 years and 2 month
  as the time from the date of the first obinutuzumab infusion to the first occurrence of molecular disease relapse
Overall survival (OS) | 3 years and 2 month
  defined as the time from the date of the initiation of the first line treatment to the death from any reason
Time to relapse/progression | 3 years and 2 month
  defined as the time from the date of the first obinutuzumab infusion to the first evidence of disease progression or relapse, as determined by the investigator using the Lugano Classification
Event-free survival (EFS) | 3 years and 2 month
  defined as the time from the date of the first obinutuzumab infusion to the first evidence of disease progression or relapse (as determined by the investigator using the Lugano Classification), death from any reason, start of the another anti-lymphoma treatment, SAE preventing continuation of the protocol treatment
Health status measured with EQ-5D from EuroQoL Group | 3 years and 2 month
  with EQ-5D from EuroQoL Group
Treatment tolerability assessment | 3 years and 2 month
  reporting of serious adverse events (SAEs), adverse events (AEs) and adverse events of special interest

CONTACTS AND LOCATIONS:
Overall Officials: Michał Szymczyk, MD, Principal Investigator — Institute of Oncology
Locations (1):
- Centrum Onkologii - Instytut im. Marii Skłodowskiej- Curie Klinika Nowotworów Układu Chłonnego, Warsaw, Poland